CLINICAL TRIAL: NCT01617213
Title: Autologous Peripheral Blood Stem Cell Transplantation and Maintenance Lenalidomide After High-dose Melphalan for Multiple Myeloma
Brief Title: Autologous Stem Cell Transplantation and Maintenance Therapy for Multiple Myeloma
Acronym: AMM-2011
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study is no longer needed as recent data have answered the primary hypotheses for this study.
Sponsor: University of Virginia (Other)
Responsible Party: Principal Investigator, Mary Laughlin, MD, Professor, Director of Stem Cell Transplant Program, University of Virginia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 16043
Record Dates: First submitted 2012-06-08; First posted 2012-06-12 (Estimated); Last update posted 2013-06-21 (Estimated); Status verified 2013-06

CONDITIONS: Multiple Myeloma
Keywords: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — Melphalan; Lenalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Maintenance Lenalidomide After Melphalan (Experimental)
  Interventions: Drug: Melphalan; Drug: Lenalidomide

INTERVENTIONS:
Drug: Melphalan — 200 mg/m2/IV
Drug: Lenalidomide — 10 mg daily continuously for the first 3 months, then increased to 15 mg daily as long as the patient tolerates the drug.

SUMMARY:
This trial will determine the feasibility and efficacy of lenalidomide as maintenance therapy in Multiple Myeloma patients treated with dose intensive chemotherapy (Melphalan 200 mg/m2) with autologous PBSC transplant.

ELIGIBILITY:
Inclusion Criteria:

* Must be 18 to 75 years of age.
* ECOG performance status of 0, 1 or 2.
* Patients who have a history of another malignant disorder are eligible, provided that they have not received active therapy for 5 years. Patients with basal cell and squamous cell skin cancers are eligible.
* Patients who are pregnant are ineligible.
* Patients must furnish written informed consent and HIPAA authorization for release of personal health information.
* Patients must be able to understand the requirements of the study, abide by the study restrictions, and agree to return for the required assessments.
* Patients must be HIV and HTLV-I,-II antibody sero-negative.
* Patients must have adequate visceral organ function

Exclusion Criteria:

* Patients are ineligible if they have received cumulative chemotherapy doses in excess of: carmustine (BCNU) 400 mg/m2, or a cumulative anthracycline exposure in excess of 550 mg/m2 Adriamycin (doxorubicin) unless the gated-pool radionuclide cardiac scan shows greater than/equal to 45% ejection fraction.
* Patients are ineligible if they are receiving any other investigational agents.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2012-04; Primary Completion 2015-04 (Estimated)

PRIMARY OUTCOMES:
Event Free Survival | 3 years
  Duration of time until patient experiences an event (recurrence, relapse or death)

SECONDARY OUTCOMES:
Disease Response | 2 years
  Number of patients that have complete and very good partial responses.
Overall survival | 4 years
  Duration of time from Day 0 until death.
Grade > 2 toxicities | 4 years
  Percent of patients experiencing one or more toxicity greater than 2.
Incidence of infections | 4 years
  Percent of patients experiencing a definite or probable viral, fungal or bacterial infection.
Treatment related Mortality | 4 years
  Number of patients that experience a death from causes other relapse or progression.

CONTACTS AND LOCATIONS:
Overall Officials: Mary J. Laughlin, MD, Principal Investigator — University of Virginia
Locations (1):
- University of Virginia, Charlottesville, Virginia, United States